CLINICAL TRIAL: NCT00630032
Title: Randomized, Open Label, Multicentric Phase III Evaluating the Benefit of a Sequential Regimen Associating FEC 100 and Ixabepilone in Adjuvant Treatment of Non Metastatic, Poor Prognosis Breast Cancer Defined as Triple-negative Tumor [HER2 Negative - ER Negative - PR Negative] or [HER2 Negative and PR Negative] Tumor; in Node Positive or Node Negative Patients.
Brief Title: Safety and Efficacy Comparison of Docetaxel and Ixabepilone in Non Metastatic Poor Prognosis Breast Cancer
Acronym: TavIx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACS08 - UC-0140/0610; PACS-08/0610 (Other: UNICANCER); 2006-006494-24 (EudraCT Number); PACS08-Tavlx (Other: UNICANCER); BMS-UNICANCER-PACS-08/0610 (Other: UNICANCER); AMGEN-UNICANCER-PACS-08/0610 (Other: UNICANCER)
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Active Comparator): 3 cycles of FEC100 (F and C, each at 500 mg/m², E 100 mg/m², every 3 weeks) followed by 3 cycles of D (100 mg/m² every 3 weeks)
  Interventions: Drug: cyclophosphamide; Drug: Docetaxel; Drug: epirubicin hydrochloride; Drug: fluorouracil
- Ixabepilone (Experimental): 3 cycles of FEC100 (F and C, each at 500 mg/m², E 100 mg/m², every 3 weeks) followed by 3 cycles of Ixabepilone (40 mg/m² every 3 weeks);
  Interventions: Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: ixabepilone

INTERVENTIONS:
Drug: cyclophosphamide — 500 mg/m² every 3 weeks
Drug: Docetaxel — 100 mg/m² every 3 weeks
  Arms: Docetaxel
Drug: epirubicin hydrochloride — 100 mg/m² every 3 weeks
Drug: fluorouracil — 500 mg/m² every 3 weeks
Drug: ixabepilone — 40 mg/m² every 3 weeks
  Arms: Ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them after surgery may kill any tumor cells remaining after surgery. It is not yet known whether docetaxel is more effective than ixabepilone when given after surgery and combination chemotherapy in treating breast cancer.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy followed by docetaxel or ixabepilone to compare how well they work in treating patients who have undergone surgery for nonmetastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the benefit from sequential administration of 3 courses of combination chemotherapy (FEC100) followed by 3 courses of ixabepilone versus docetaxel on the 5-year disease-free survival of women with nonmetastatic, poor-prognosis breast cancer.

Secondary

* To compare the 5-year distant metastasis-free survival.
* To compare the 5-year event-free survival.
* To compare the 5-year overall survival.
* To compare the safety profiles for the two chemotherapy regimens.
* To identify and/or validate predictive-gene expression profiles of clinical response/resistance to the two treatment regimens.
* To bank frozen and fixed tumor and frozen serum prospectively for future translational studies in both genomics and proteomics (transcriptome and proteome analyses, tissue array analyses).
* To compare the cost-effectiveness of these 2 regimens.
* To compare the quality-of-life of patients treated with these 2 regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, menopausal status (pre- vs post-menopausal), and tumor hormone-receptor status (triple-negative vs progesterone-receptor negative, HER negative, and estrogen-receptor [ER] positive). Patients are randomized to 1 of 2 treatment arms.

* Docetaxel Arm: Patients receive epirubicin hydrochloride IV, fluorouracil IV, and cyclophosphamide IV every 3 weeks in courses 1-3 and docetaxel IV alone every 3 weeks in courses 4-6.
* Ixabepilone Arm: Patients receive treatment in courses 1-3 as in arm I and ixabepilone IV alone every 3 weeks in courses 4-6.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients also complete a quality of life questionnaire periodically.

After completion of study treatment, patients are followed periodically for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically proven invasive unilateral breast cancer (regardless of the type)

  * Initial clinical condition compatible with complete initial resection
  * No residual macro or microscopic tumor after surgical excision
* Node-positive disease (i.e., positive sentinel node or positive axillary clearance) (N+) or node-negative disease (-) meeting the following criteria :

  * Stage II or III disease
  * pT >20 mm (T1-4)
* Patients must meet 1 of the following hormone-receptor criteria:

  * Node-positive patients: triple-negative* tumor (HER2 negative, estrogen-receptor [ER] negative, and progesterone receptor [PR] negative) OR double-negative (HER2 negative, PR negative, and ER+)
  * Node-negative patients: triple-negative* tumor only
* NOTE: *Hormone-receptor negativity is defined as ER <10% and PR <10% by IHC and HER2 negativity is defined as IHC 0-1+ OR IHC 2+ and FISH or CISH negative
* Must be able to begin chemotherapy no later than day 49 after the initial surgery

Exclusion criteria:

* Clinically or radiologically detectable metastases (M0)
* Bilateral breast cancer or contralateral ductal carcinoma in situ
* Any metastatic impairment, including homolateral subclavicular node involvement, regardless of its type
* Any tumor ≥T4a (cutaneous invasion, deep adherence, inflammatory breast cancer)
* HER 2 overexpression defined as IHC 3+ OR IHC 2+ and FISH or CISH positive
* Any clinically or radiologically suspect and non-explored damage to the contralateral breast

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Pre- or postmenopausal
* ECOG performance status 0-1
* Peripheral neuropathy ≤grade 1
* Neutrophil count ≥2,000/mm³
* Platelet count ≥100,000/mm³
* Hemoglobin >9 g/dL
* AST and ALT ≤1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤2.5 times ULN
* Total bilirubin ≤1.0 times ULN
* Serum creatinine ≤1.5 times ULN
* LVEF ≥50% by MUGA scan or echocardiography
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 8 weeks after completion of study treatment

Exclusion criteria:

* Previous cancer (except cutaneous baso-cellular epithelioma or uterine peripheral epithelioma) in the preceding 5 years, including invasive contralateral breast cancer
* Patients with any other concurrent severe and/or uncontrolled medical disease or infection that could compromise participation in the study
* Clinically significant cardiovascular disease within the past 6 months including any of the following:

  * Unstable angina
  * Congestive heart failure
  * Uncontrolled hypertension (i.e., blood pressure >150/90 mm Hg)
  * Myocardial infarction
  * Cerebral vascular accidents
* Known prior severe hypersensitivity reactions to agents containing Cremophor EL
* Patients with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Patients deprived of liberty or placed under the authority of a tutor

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior minor surgery (excluding breast biopsy) and adequately recovered
* At least 3 weeks since prior major surgery and adequately recovered
* No prior chemotherapy, hormonal therapy, or radiotherapy
* More than 72 hours since prior and no concurrent treatment with any of the following strong inhibitors of CYP3A4:

  * Amiodarone
  * Clarithromycin
  * Amprenavir
  * Delavirdine
  * Voriconazole
  * Erythromycin
  * Fluconazole
  * Itraconazole
  * Ketoconazole
  * Indinavir
  * Nelfinavir
  * Ritonavir
  * Saquinavir
* No concurrent participation in another therapeutic trial involving an experimental drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Campone, MD, Principal Investigator — ICO Centre Regional Rene Gauducheau
Locations (86):
- United States (17):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Southeast Nebraska Hematology Oncology Consultants at Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Oncology Associates at Rapid City Regional Hospital, Rapid City, South Dakota
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Centre de Sante des Fagnes, Chimay
  - Centre Hospitalier Hutois, Huy
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - CHR - Clinique Saint Joseph - Hopital de Warqueguies, Mons
  - Clinique Saint-Pierre, Ottignies
  - Clinique Universitaire De Mont-Godinne, Yvoir
- France (62):
  - Clinique Claude Bernard, Albi
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Blois, Blois
  - Institut Bergonie, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier de Fleyriat, Bourg-en-Bresse
  - CHU Hopital A. Morvan, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Regional de Chambery, Chambéry
  - Centre Hospitalier de Chateaubriant, Châteaubriant
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique des Cedres, Cornebarrieu
  - Hopital Intercommunal De Creteil, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Clinique Claude Bernard, Ermont
  - Hopital Jean Monnet, Épinal
  - Hopital Andre Mignot, Le Chesnay
  - CMC Les Ormeaux, Le Havre
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre Leon Berard, Lyon
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Clinique Claude Bernard, Metz
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Clinique du Pont de Chaume, Montauban
  - Centre Hospitalier Intercommunal Le Raincy - Montfermeil, Montfermeil
  - Centre Hospitalier de Montlucon, Montluçon
  - Centre Hospitalier, Mulhouse
  - Clinique D'Occitanie, Muret
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Clinique De Valdegour, Nîmes
  - Hopital Saint Michel, Paris
  - Institut Curie Hopital, Paris
  - Centre Hospitalier - Pau, Pau
  - Centre Hospitalier de Perpignan, Perpignan
  - Polyclinique Francheville, Périgueux
  - Institut Jean Godinot, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier de Rodez, Rodez
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Regional Rene Gauducheau, Saint-Herblain
  - Clinique de l'Union, Saint-Jean
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Clinique de l'Orangerie, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Polyclinique de L'Ormeau, Tarbes
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Institut Claudius Regaud, Toulouse
  - Clinique Du Parc, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Centre d'Oncologie Saint-Yves, Vannes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- See also: Abstract primary endpoint results — https://www.ncbi.nlm.nih.gov/pubmed/30267987

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel: 3 cycles of FEC100 (F and C, each at 500 mg/m², E 100 mg/m², every 3 weeks) followed by 3 cycles of D (100 mg/m² every 3 weeks)
  Cyclophosphamide: 500 mg/m² every 3 weeks Docetaxel: 100 mg/m² every 3 weeks Epirubicin hydrochloride: 100 mg/m² every 3 weeks Fluorouracil: 500 mg/m² every 3 weeks
- Ixabepilone: 3 cycles of FEC100 (F and C, each at 500 mg/m², E 100 mg/m², every 3 weeks) followed by 3 cycles of Ixabepilone (40 mg/m² every 3 weeks);
  Cyclophosphamide: 500 mg/m² every 3 weeks Epirubicin hydrochloride: 100 mg/m² every 3 weeks Fluorouracil: 500 mg/m² every 3 weeks Ixabepilone: 40 mg/m² every 3 weeks
Period: Overall Study
Arm/Group | Docetaxel | Ixabepilone
Started | 398 | 364
Completed | 308 | 269
Not Completed | 90 | 95
Not completed — Death | 55 | 49
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 18 | 31
Not completed — Protocol Violation | 1 | 0
Not completed — Patient has moved | 1 | 1
Not completed — Disease progression | 1 | 1
Not completed — End of monitoring in US centers | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel | Ixabepilone | Total
Number analyzed (Participants) | 398 | 364 | 762
Age, Continuous [Median (Full Range); unit: years] | 53.5 [24 to 71] | 53 [26 to 71] | 53 [24 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 398 | 364 | 762
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 92 | 74 | 166
  United States | 12 | 13 | 25
  France | 294 | 277 | 571

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease-free Survival (DFS)
Description: DFS is defined as the interval between the date of randomization and the date of breast cancer relapse (local, regional or distant) or the date of invasive contralateral breast cancer or death from any cause, whichever occurs first
Time Frame: At 5 years
Population: The DFS was analyzed in the intention-to-treat population: All subjects randomized to a treatment arm with or without treatment (N=762).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 398 | 364
Percentage of participants | 78.97 [74.53 to 82.73] | 83.37 [79.06 to 86.87]
Statistical Analysis 1: Comparison: Docetaxel vs Ixabepilone; Test type: Superiority; p = 0.175, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.10]

2. Secondary Outcome: Number of Disease-free Survival Events for Triple-negative Subgroup
Description: DFS is defined as the interval between the date of randomization and the date of breast cancer relapse (local, regional or distant) or the date of invasive contralateral breast cancer or death from any cause, whichever occurs first in participants with triple negative breast cancer only.
Time Frame: At 5 years
Population: The DFS for triple-negative subgroup was analyzed in all triple negative breast cancer participants randomized to a treatment arm with or without treatment (N=586).
Measure: Number; unit: Events
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 307 | 279
Events | 69 | 50
Statistical Analysis 1: Comparison: Docetaxel; Test type: Superiority; p = 0.1687, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.53 to 1.11]

3. Secondary Outcome: Number of Disease-free Survival Events for ER+/PR-/HER2- Subgroup
Description: DFS is defined as the interval between the date of randomization and the date of breast cancer relapse (local, regional or distant) or the date of invasive contralateral breast cancer or death from any cause, whichever occurs first in participants with ER+/PR-/HER2- breast cancer only.
Time Frame: At 5 years
Population: The DFS for ER+/PR-/HER2- subgroup was analyzed in all ER+/PR-/HER2- breast cancer participants randomized to a treatment arm with or without treatment (N=167).
Measure: Number; unit: Events
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 85 | 82
Events | 21 | 17
Statistical Analysis 1: Comparison: Docetaxel vs Ixabepilone; Test type: Superiority; p = 0.6502, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.45 to 1.63]

4. Secondary Outcome: Number of Distant Metastasis-free Survival Events for the Whole Population
Description: The distant metastases-free survival is the length of time during and after the treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body.
Time Frame: At 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 398 | 364
Events | 82.3 [78.1 to 85.8] | 87.7 [83.8 to 90.7]
Statistical Analysis 1: Comparison: Docetaxel vs Ixabepilone; Test type: Superiority; p = 0.0665, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.49 to 1.02]

5. Secondary Outcome: Number of Event-free Survival
Description: The Event-free Survival is defined as the interval between the date of randomization and the date of breast cancer relapse (local, regional or distant) or the date of invasive contralateral breast cancer or the date of second neoplasia, or the date of death from any cause, whichever occurs first.
Time Frame: At 5 years
Measure: Number (95% Confidence Interval); unit: Events
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 398 | 364
Events | 77.46 [72.94 to 81.32] | 81.53 [77.05 to 85.22]
Statistical Analysis 1: Comparison: Docetaxel vs Ixabepilone; Test type: Superiority; p = 0.148, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.59 to 1.08]

6. Secondary Outcome: Overall Survival
Description: The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Time Frame: At 5 years
Population: The OS was analyzed in the intention-to-treat population: All subjects randomized to a treatment arm with or without treatment (N=762).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel | Ixabepilone
Number analyzed (Participants) | 398 | 364
percentage of participants | 87.00 [83.13 to 90.03] | 87.60 [83.64 to 90.66]
Statistical Analysis 1: Comparison: Docetaxel vs Ixabepilone; Test type: Superiority; p = 0.8968, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.67 to 1.42]

ADVERSE EVENTS:
Time Frame: Throughtout the study, up to 5 years
Arm/Group | Docetaxel | Ixabepilone
All-Cause Mortality (participants affected / at risk) | 58/398 | 51/364
Serious Adverse Events (participants affected / at risk) | 207/398 | 158/364
Other Adverse Events (participants affected / at risk) | 398/398 | 364/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=398) | Ixabepilone (N=364)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Aplasia bone marrow (Blood and lymphatic system disorders) | 1 | 1
Febrile aplasia (Blood and lymphatic system disorders) | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 56 | 27
Lymphocele (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 141 | 95
Auricular fibrillation (Cardiac disorders) | 1 | 0
Non ST segment elevation acute coronary syndrome (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Cataract (left) (Eye disorders) | 1 | 0
Eye infection (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Crohn's enteritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction complicating hernia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Epigastralgia (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 5 | 1
Mucositis (General disorders) | 2 | 3
Pain (General disorders) | 1 | 0
Hepatic dysfunction NOS (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 1
Allergy (Immune system disorders) | 0 | 3
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 3
Device complication (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Infection injection site (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Abscess soft tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of cardia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloid leukemia, acute (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoma of tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreas cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Pain nerve (Nervous system disorders) | 1 | 0
Schwannoma (Nervous system disorders) | 1 | 0
Cerebral hypoperfusion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 10
Sensory neuropathy (Nervous system disorders) | 1 | 4
Melancholia (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Infection urinary tract (Renal and urinary disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Exfoliative dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Fingernail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Recall phenomenon (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Allergic skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Device implant NOS (Surgical and medical procedures) | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1
Pulmonary embolism (Vascular disorders) | 1 | 2
Jugular vein thrombosis (Vascular disorders) | 1 | 1
Thrombosis cerebral vein (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (N=398) | Ixabepilone (N=364)
Anemia (Blood and lymphatic system disorders) | 325 | 287
Febrile neutropenia (Blood and lymphatic system disorders) | 67 | 52
neutropenia (Blood and lymphatic system disorders) | 328 | 314
Thrombopenia (Blood and lymphatic system disorders) | 72 | 87
Alopecia (Skin and subcutaneous tissue disorders) | 317 | 307
Cardiovascular disorder (Cardiac disorders) | 31 | 45
Cutaneous (Skin and subcutaneous tissue disorders) | 158 | 113
Edema (Cardiac disorders) | 67 | 59
Fever (General disorders) | 83 | 71
Hepatic (Hepatobiliary disorders) | 13 | 43
Infection (Infections and infestations) | 120 | 123
Mucitis (Vascular disorders) | 210 | 185
Nausea (Gastrointestinal disorders) | 325 | 295
Neurotoxicity peripheral (Nervous system disorders) | 33 | 59
Sensory neurotoxicity (Nervous system disorders) | 99 | 164
Nail disorder (Skin and subcutaneous tissue disorders) | 100 | 73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT00630032/Prot_SAP_000.pdf